CLINICAL TRIAL: NCT05916989
Title: Stimulant Use and Methylation in HIV
Status: Completed | Type: Observational
Sponsor: Florida International University (Other)
Collaborators: New York University (Other); Northwestern University (Other); University of California, San Francisco (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Carrico, PhD, Professor and Chair, Florida International University
Other Study IDs: 20180865; R01DA033854 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections; Methamphetamine-dependence; Methamphetamine Abuse
Keywords: HIV; Methamphetamine; Methylation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Leukocyte DNA Samples: Leukocyte DNA specimens extracted from participants enrolled in a completed NIH funded trial will be examined to determine if prior exposure to different behavioral interventions modifies DNA methylation patterns over 6 months.

SUMMARY:
This study will leverage extracted leukocyte DNA specimens from a completed NIH-funded project to examine the efficacy of a behavioral intervention model that reduced stimulant use on DNA methylation over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Documentation of HIV-positive serostatus
* Speak English
* Biological verification of recent methamphetamine use
* Completion of at least three contingency management (CM) visits
* Self reported anal sex with a man in the past 12 months

Exclusion Criteria:

* Inability to provide informed consent, evidenced by cognitive impairment
* HIV negative serostatus

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sexual Minority Men - gay, bisexual, and other men who have sex with men.
Study Population: Sexual minority men with HIV who use methamphetamine residing in the San Francisco Bay Area.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Neuroimmune Signaling | 6 Months
  Decreased methylation of genes for genes relevant to neuroimmune signaling such as beta-2 (β2) adrenergic (i.e., ADRB2), glucocorticoid (i.e., NR3C1 and FKBP5), and oxytocin (i.e., OXTR) receptors as well as brain-derived neurotrophic factor (BDNF) promoters.

SECONDARY OUTCOMES:
DNA Methylation Pathways | 6 Months
  Pathway Analyses examining alterations in methylation patterns relevant to immune and neural function.
Immune Dysfunction | 6 Month
  Soluble makers of monocyte activation such as soluble CD14 (sCD14) and inflammation such as soluble Tumor Necrosis Factor - Alpha Receptors I and II (sTNF-aRI and sTNF-aRII)
Dysregulated Metabolism of Amino Acid Precursors for Neurotransmitters measured via high-performance liquid chromatography (HPLC) | 6 Months
  Using HPLC, higher kynurenine/tryptophan (K/T) ratio indexes catabolism of tryptophan into kynurenine and other downstream catabolites versus serotonin over 6 months. Using HPLC, the phenylalanine/tyrosine ratio reflects decreased metabolism of tyrosine into catecholamines such as dopamine over 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Carrico, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No